CLINICAL TRIAL: NCT01382108
Title: Meibography and Tear Scan Using the Oculus Keratograph 4
Acronym: KITCHENER
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, Centre for Contact Lens Research, Lyndon Jones, PhD, University of Waterloo
Other Study IDs: P/374/11/CCLR
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-10

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal participants
- Meibomian Gland Dysfunction

SUMMARY:
The purpose of this study is to look at both the meibomian glands and the tear film using a new clinical instrument marketed in Canada which was recently acquired by the Centre for Contact Lens Research. These will be compared between two groups of individuals, one group with visible meibomian gland dysfunction (MGD) and one group of individuals with normal meibomian gland appearance. The hypothesis is that there will be a difference between normal individuals and individuals with MGD with respect to the appearance of the meibomian glands and certain tear film attributes.

DETAILED DESCRIPTION:
Meibomian gland dysfunction (MGD) is a common clinical condition and a major cause of evaporative dry eye with associated discomfort, visual disturbance and contact lens intolerance. In MGD, meibum is often abnormal, progressively changing in color from clear to yellow and in consistency from liquid to thick and toothpaste-like. Evaluation of the meibomian glands (MG) and lipid layer is vital. In a typical clinical setting, lid and lid margin evaluation is often performed via slitlamp biomicroscopy; however, the structure of the meibomian glands is often not clearly visualized when a slit lamp is used in isolation. Trans-illumination of the lids is necessary to clearly view these glands.

To date, infrared meibography has been the only method available for the assessment of meibomian gland structure. It is primarily regarded as a laboratory-specific procedure for meibomian gland drop out assessment in people suffering from MGD. Recently, the Keratograph 4 was released by OCULUS (Wetzlar, Germany). In addition to corneal and contact lens assessment features, the Keratograph 4 offers a tear film (TF) scan module able to objectively assess tear break-up time (TBUT) with a colour coded map highlighting the regions of tear break up. High-resolution images of tear meniscus can also be obtained and used for subjective assessment of tear meniscus height (TMH) with the help of built-in software. Preliminary research at the Centre for Contact Lens Research has demonstrated its ability to capture meibography images of the upper and lower lids.

The objectives of this study are to collect meibography, TBUT and TMH data using the Keratograph 4 in normal participants (no MGD) and participants with MGD and to compare these between the two groups and before and after the use of a meibomian gland evaluator. The primary outcome variables are meibography images, TBUT and TMH.

The study hypothesis is that here will be a difference between normal participants and participants with MGD, with respect to meibography images (MG drop out), TBUT measurements (area and time of break up) and TMH measurements.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer
* Has read and signed an information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Has had an ocular examination in the last two years
* Clinical criteria defining non-dry eye (controls) for study inclusion (Group 1):

  1. Composite symptom score of ≤ 12 on the OSDI questionnaire
  2. Meibum secretion quality score of 0 (grade 0-3) at the central eight meibomian glands of the lower lid, in both eyes. Secretion quality score (grade 0-3):

Grade 0 = normal, clear oil expressed (i.e., cooking oil appearance) Grade 1= opaque, diffusely turbid, normal viscosity Grade 2 = opaque, increased viscosity Grade 3 = inspissated (i.e., toothpaste-like appearance) or no expressed material Clinical criteria defining MGD dry eye for study inclusion (Group 2):

1. Composite symptom score of ≥ 13 on the OSDI questionnaire
2. Meibum secretion quality score ≥ 1.0 (grade 0-3) at the central eight meibomian glands of the lower lid, in both eyes. Secretion quality score (grade 0-3):

Grade 0 = normal, clear oil expressed (i.e., cooking oil appearance) Grade 1 = opaque, diffusely turbid, normal viscosity Grade 2 = opaque, increased viscosity Grade 3 = inspissated (i.e., toothpaste-like appearance) or no expressed material

Exclusion Criteria:

* Is a current contact lens wearer
* Has any ocular disease
* Is using any topical medications that may affect ocular health
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Non-contact lens wearers will be recruited using CCLR records and advertising approved by the UW Office of Research Ethics
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 non-contact lens wearers were recruited using CCLR records
Groups:
- Normal Participants: Participants without Meibomian Gland Dysfunction
- Meibomian Gland Dysfunction: Participants with Meibomian Gland Dysfunction
Period: Overall Study
Arm/Group | Normal Participants | Meibomian Gland Dysfunction
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Participants | Meibomian Gland Dysfunction | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 31
  >=65 years | 3 | 5 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (6.1) | 59.5 (10.8) | 58.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Meibomium Gland Dropout Score - Evidence of Meibomian Gland Dysfunction (MGD) Confirmed by Meibograhpy Imaging Using the Keratograph 4 Measured on a Subjective Grading Scale (0-3) (Summing the Score for the Upper and Lower Lids for a Final Scale of 0-6)
Description: Assessments will be made in normal participants (no MGD) and participants with MGD and compared between the two groups at baseline and after the use of a meibomian gland evaluator.
  The meibomium gland dropout score subjective grading scale:
  0 = no loss of mebomium glands
  1. = area of meibomium gland loss less than 33%
  2. = area of meibomium gland loss between 33% and 67%
  3. = area of meibomium gland loss more than 67%.
Time Frame: Before and after the use of a meibomian gland evaluator. Assessments will be separated by a period of at least 10 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Participants | Meibomian Gland Dysfunction
Number analyzed (Participants) | 20 | 19
units on a scale
  Subjective grading (0-6) (baseline) | 1.3 (1.0) | 3.1 (1.1)
  Subjective grading (0-6) (after 10 minutes) | 1.3 (1.0) | 3.1 (1.1)

2. Primary Outcome: Tear Breakup Time (TBUT). The Time Taken, in Seconds, for the Tear Film to Break up on the Surface of the Cornea.
Description: Measurements will be made in normal participants (no MGD) and participants with MGD and compared between the two groups at baseline and after the use of a meibomian gland evaluator.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Normal Participants | Meibomian Gland Dysfunction
Number analyzed (Participants) | 20 | 19
seconds
  TBUT (baseline) | 9.0 (6.6) | 6.7 (6.8)
  TBUT (after 10 minutes) | 6.8 (6.1) | 7.6 (6.8)

3. Primary Outcome: Tear Meniscus Height (TMH). The Height of the Tear Film Meniscus at the Eyelid Margin.
Description: Assessments will be made in normal participants (no MGD) and participants with MGD and compared between the two groups at baseline and after the use of a meibomian gland evaluator.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Normal Participants | Meibomian Gland Dysfunction
Number analyzed (Participants) | 20 | 19
mm
  TMH (baseline) | 0.2 (0.1) | 0.2 (0.1)
  TMH (after 10 minutes) | 0.2 (0.1) | 0.2 (0.1)

ADVERSE EVENTS:
Arm/Group | Normal Participants | Meibomian Gland Dysfunction
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes